CLINICAL TRIAL: NCT02768090
Title: Proteomic Analysis of Sweat in Cutaneous Inflammatory and Neoplastic Conditions
Brief Title: Proteomic Analysis of Sweat in Cutaneous Conditions
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study Period Ended / Not Completed
Sponsor: Larkin Community Hospital (Other)
Collaborators: George Mason University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LCH-1-012016
Record Dates: First submitted 2016-05-09; First posted 2016-05-11 (Estimated); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Application Site Perspiration
MeSH Terms: interventions — Transdermal Patch

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Skin Patch (Experimental): Sweat will be collected from inflammatory and neoplastic skin lesions with an FDA approved diagnostic skin patch for analysis with mass spectrometry
  Interventions: Device: Skin Patch

INTERVENTIONS:
Device: Skin Patch — Sweat will be collected by applying a diagnostic skin patch to inflammatory and neoplastic cutaneous lesions for proteomic analysis with mass spectrometry.

SUMMARY:
This study will investigate a new diagnostic technology in order to expand current understanding of inflammatory and neoplastic cutaneous disease processes such as eczema, psoriasis, granuloma annulare, cutaneous lymphoma, squamous cell carcinoma, basal cell carcinoma and melanoma. Protein fragments found in sweat will be collected using a diagnostic skin patch and analyzed with mass spectrometry. The goal of this study is to identify specific protein fragment biomarkers that may further current understanding of cutaneous diseases. The protein expression patterns derived from sweat will be compared to conventional histopathologic, immunohistochemical, flow cytometry, in-situ hybridization, polymerase chain reaction, and mass spectrometry analyses of cutaneous biopsy specimens. The insight gained from this research will be used to promote advances in disease prevention and early diagnosis, identify prognostic indicators and new therapeutic targets.

DETAILED DESCRIPTION:
The investigators propose a novel technology to be used at the bedside or in the field: an FDA approved diagnostic skin patch which harvests, concentrates, and stabilizes a panel of protein fragments derived from skin transudate or sweat. While drug delivery patches are routinely used, the technology proposed here has exactly the opposite function: the harvesting of diagnostic markers using novel affinity bait nanoparticles, bound within an adhesive skin patch. The proposed technology may overcome all major physiological barriers that have prevented the use of this biologic fluid for diagnostic testing. Sweat disease protein fragments are subject to rapid degradation due to proteases present in sweat and normal skin bacterial flora, and exist in extremely low abundance, far below the detection sensitivity of standard analysis platforms. Harvesting hydrogel nanoparticles are engineered with chemical high affinity baits so that they sequester the low abundance target analytes, and protect them from degradation indefinitely. Once applied to the skin, the nanoparticles in the patch harvest minute by minute, and protect from degradation, all candidate analytes in the sweat underneath the patch. The core shell bait nanoparticles are a completely novel technology that can amplify the sensitivity of protein fragment detection by 100 fold. No other technology exists that has a similar yield, concentration ability, and stabilization function. Once the collection is complete, the patch will be mailed to the diagnostic lab at room temperature. Upon receipt, the nanoparticle-captured analytes of interest can be eluted from the patch for routine measurement using any platform. Feasibility studies have demonstrated virtually 100 percent capture and 100 percent elution yield of low abundance interleukins in model sweat solutions. The investigators will collect sweat from healthy volunteers under Institutional Review Board approval. Mass spectrometry will be used to discover novel sweat protein fragments that have been concentrated and preserved in the patch. Low abundance labile protein fragments harvested from the nanoparticles will be measured by clinical immunoassays to verify sensitivity and precision. Data gathered from this study will be used to develop a foundation for sweat protein fragment testing of cutaneous disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients who present with an inflammatory or neoplastic skin condition at approved study locations will be screened for eligibility. All patients > 18 years of age with a suspected cutaneous malignancy. Face and body sites will be included. No maximum number of areas are set and will depend on the areas deemed clinical appropriate and necessary for accurate diagnosis

Exclusion Criteria:

* Exclusion criteria include patients enrolled in investigational drug clinical trials, patients who received or currently receive systemic chemotherapy, pregnancy, persons < 18 years of age, and persons whom are unable to consent to medical procedures themselves.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-02-25 (Actual); Primary Completion 2017-01-30 (Actual); Study Completion 2017-01-30 (Actual)

PRIMARY OUTCOMES:
Analysis of perspired protein fragments in cutaneous diseases | 1 year
  Mass spectrometry will be used to identify protein fragments from sweat collected from a skin patch that will be applied directly to skin lesions of eczema, psoriasis, granuloma annulare, cutaneous lymphoma, basal cell carcinoma, squamous cell carcinoma and melanoma. These protein fragments will be compared to protein fragments perspired from normal skin in order to look for signature patterns of expression that correlate to each disease entity. Low abundance labile sweat protein fragments harvested from the nanoparticles will be measured by clinical immunoassays to verify sensitivity and precision.

CONTACTS AND LOCATIONS:
Overall Officials: Laszlo Karai, MD, PhD, Principal Investigator — Larkin Community Hospital; Edwardo Weiss, MD, Study Director — Larkin Community Hospital; Bertha Baum, DO, Study Chair — Larkin Community Hospital
Locations (1):
- Hollywood Dermatology, Hollywood, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fredolini C, Meani F, Reeder KA, Rucker S, Patanarut A, Botterell PJ, Bishop B, Longo C, Espina V, Petricoin EF 3rd, Liotta LA, Luchini A. Concentration and Preservation of Very Low Abundance Biomarkers in Urine, such as Human Growth Hormone (hGH), by Cibacron Blue F3G-A Loaded Hydrogel Particles. Nano Res. 2008 Dec;1(6):502-518. doi: 10.1007/s12274-008-8054-z. PMID 20467576
- [Background] Longo C, Patanarut A, George T, Bishop B, Zhou W, Fredolini C, Ross MM, Espina V, Pellacani G, Petricoin EF 3rd, Liotta LA, Luchini A. Core-shell hydrogel particles harvest, concentrate and preserve labile low abundance biomarkers. PLoS One. 2009;4(3):e4763. doi: 10.1371/journal.pone.0004763. Epub 2009 Mar 10. PMID 19274087